CLINICAL TRIAL: NCT07361094
Title: An Exploratory Clinical Study to Evaluate the Safety and Efficacy of Autologous CD19-BCMA Dual-Target Chimeric Antigen Receptor T-Cell Therapy in Patients With Relapsed or Refractory Autoimmune Diseases
Brief Title: Autologous CD19/BCMA Dual-Target CAR-T for Relapsed/Refractory Autoimmune Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Boren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJBR-2025-AID-001
Record Dates: First submitted 2026-01-04; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory Systemic Lupus Erythematosus; Relapsed/Refractory Systemic Sclerosis; Relapsed/Refractory Idiopathic Inflammatory Myopathies; Relapsed/Refractory sjögren's Syndrome; Relapsed/Refractory Autoimmune Hemolytic Anemia; Relapsed/Refractory Multiple Sclerosis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Scleroderma, Systemic; Myositis; Sjogren's Syndrome; Anemia, Hemolytic, Autoimmune; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous CD19-BCMA Dual-Target CAR T-Cell Therapy (Fixed Dose) (Experimental): The study uses a fixed dose of 1 × 10⁶ CAR-T cells per kilogram of body weight for infusion, followed by a 24-month follow-up period after cell infusion to evaluate safety and efficacy.
  Interventions: Drug: Autologous CD19-BCMA Dual-Target CAR T-Cell Therapy

INTERVENTIONS:
Drug: Autologous CD19-BCMA Dual-Target CAR T-Cell Therapy — Autologous CD19-BCMA dual-target CAR T-cell therapy is a personalized cell-based immunotherapy manufactured from each participant's own peripheral blood T lymphocytes. Following leukapheresis, autologous T cells are genetically modified ex vivo to express a chimeric antigen receptor targeting both CD19 and B-cell maturation antigen (BCMA), enabling recognition and elimination of B-lineage cells and antibody-producing plasma cells implicated in autoimmune disease pathogenesis. The modified T cells are expanded under controlled conditions and administered as a single intravenous infusion after lymphodepleting conditioning. This dual-target CAR-T approach is intended to provide broad and sustained depletion of pathogenic B-cell populations and to promote immune system rebalancing in patients with relapsed or refractory autoimmune diseases.

SUMMARY:
Autoimmune diseases occur when the immune system mistakenly attacks the body's own tissues, leading to chronic inflammation and damage to organs such as the kidneys, lungs, muscles, nerves, or blood cells. Although many treatments are available, some patients do not respond adequately or experience repeated disease flares despite long-term therapy. New treatment approaches are therefore needed for patients with relapsed or refractory autoimmune diseases. This study is an exploratory clinical trial designed to evaluate the safety and potential benefits of a novel cell-based therapy called autologous CD19-BCMA dual-target CAR T-cell therapy. This treatment uses a patient's own immune cells, which are collected from the blood, modified in the laboratory to recognize specific immune cells involved in autoimmune disease, and then infused back into the patient. The study includes adult patients with certain relapsed or refractory autoimmune diseases, such as systemic lupus erythematosus, systemic sclerosis, inflammatory muscle diseases, Sjögren's syndrome, autoimmune hemolytic anemia, and multiple sclerosis. After cell collection and preparative treatment, participants will receive a single infusion of the investigational CAR T-cell therapy and will be closely monitored for safety. The main purpose of this study is to better understand the safety of this treatment, including possible side effects. The study will also explore how the disease responds to treatment over time. Participants will be followed for up to two years after treatment to assess safety and clinical outcomes. The results of this study may help researchers better understand whether this type of cell therapy could be a feasible treatment option for patients with difficult-to-treat autoimmune diseases in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years (inclusive), of any sex.
2. Patients with failure of prior single-target CD19 or BCMA therapy, with a washout period of at least 6 months since the last treatment.
3. Disease-specific criteria for different indications:

3.1 Relapsed/Refractory Moderate-to-Severe Systemic Lupus Erythematosus (SLE)

Participants must meet all of the following:

1. Diagnosis of SLE according to the 2019 EULAR/ACR Classification Criteria for Systemic Lupus Erythematosus.
2. At screening, positive antinuclear antibody (ANA) (titer ≥1:80), and/or positive anti-dsDNA antibody, and/or positive anti-Sm antibody.
3. Moderate-to-severe disease activity defined as: SLEDAI-2000 score ≥8 at screening; if hypocomplementemia and/or anti-dsDNA antibody contribute to the score, the clinical SLEDAI-2000 score (excluding low complement and/or anti-dsDNA) must be ≥6.
4. A documented history of at least 6 months of stable standard-of-care therapy for SLE prior to screening, with active disease for at least 2 months before screening. Standard therapy includes stable use (alone or in combination) of one or more of the following: glucocorticoids (≤20 mg/day prednisone or equivalent), antimalarial drugs (hydroxychloroquine ≤400 mg/day; chloroquine ≤500 mg/day), nonsteroidal anti-inflammatory drugs (NSAIDs), biologic agents (rituximab, belimumab, telitacicept), and other immunosuppressive or immunomodulatory agents including mycophenolate mofetil (≤2 g/day), azathioprine (≤2 mg/kg/day), methotrexate (≤20 mg/week), etc.

3.2 Relapsed/Refractory Systemic Sclerosis (SSc)

Participants must meet all of the following:

1. Diagnosis of SSc according to the 2013 EULAR/ACR Classification Criteria for Systemic Sclerosis.
2. Diffuse cutaneous SSc as defined by LeRoy et al. (1988), characterized by extensive skin fibrosis involving areas proximal to the elbows and/or knees.
3. Presence of interstitial lung disease (ILD) at screening, with forced vital capacity (FVC) 45-70% predicted, or diffusing capacity for carbon monoxide (DLCO) 40-70% predicted.
4. Relapsed/refractory disease defined as inadequate response to prior standard therapy or relapse after remission. Standard therapy includes glucocorticoids, cyclophosphamide, and at least one immunosuppressive or immunomodulatory agent administered for ≥6 months (e.g., azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, rituximab, belimumab, telitacicept).
5. Evidence of active disease, defined by at least one of the following: (a) progressive skin involvement at screening with an increase in modified Rodnan skin score (mRSS) ≥10% within the past 6 months; (b) evidence of active ILD, including newly diagnosed ILD within the past 6 months, or (in patients with pre-existing ILD) a decline in FVC ≥10%, or a decline in FVC ≥5% accompanied by a decline in DLCO ≥15% within the past 6 months.

   3.3 Relapsed/Refractory Idiopathic Inflammatory Myopathies (IIM)

   Participants must meet all of the following:

(1) Diagnosis of IIM with a probability ≥55% according to the 2017 EULAR/ACR Classification Criteria for IIM, and classified as dermatomyositis (DM), polymyositis (PM), or immune-mediated necrotizing myopathy (IMNM).

(2) Active or severe disease defined as: (a) Manual Muscle Testing-8 (MMT-8) score ≤141 (total score 150); and (b) at least two of the following abnormal core set measures: patient global disease activity VAS ≥2 (0-10 scale); physician global disease activity VAS ≥2 (0-10 scale); physician global extramuscular disease activity VAS ≥2 (0-10 scale); Health Assessment Questionnaire Disability Index (HAQ-DI) ≥0.25 (0-3 scale); at least one muscle enzyme level >1.5 × upper limit of normal (ULN).

3.4 Relapsed/Refractory Sjögren's Syndrome (SS)

Participants must meet all of the following:

1. Diagnosis of SS according to the 2016 EULAR/ACR Classification Criteria for Sjögren's Syndrome.
2. Positive anti-Ro/SSA antibody at screening.
3. Salivary flow rate at screening: stimulated whole salivary flow ≥0.05 mL/min, or unstimulated whole salivary flow ≥0.01 mL/min.
4. Active disease defined as ESSDAI score ≥5. 3.5 Relapsed/Refractory Autoimmune Hemolytic Anemia (AIHA)

   Participants must meet all of the following:

(1) Diagnosis consistent with the Chinese Guidelines for the Diagnosis and Treatment of Adult Autoimmune Hemolytic Anemia (2023 Edition).

(2) Evidence of hemolysis, including: anemia based on hemoglobin level; reduced haptoglobin (<250 mg/L), elevated total bilirubin (≥17.1 μmol/L, predominantly indirect), elevated lactate dehydrogenase (LDH), and reticulocyte percentage >4% or absolute reticulocyte count >120 × 10^9/L; and detection of red blood cell autoantibodies.

(3) Relapsed/refractory disease defined as inadequate response, intolerance, contraindication, or relapse after ≥3 months of treatment with glucocorticoids combined with at least one immunosuppressive agent (e.g., cyclophosphamide, azathioprine, vinca alkaloids, calcineurin inhibitors, mycophenolate mofetil) and/or rituximab.

3.6 Relapsed/Refractory Multiple Sclerosis (MS)

Participants must meet all of the following:

(1) Diagnosis of MS according to the Chinese Guidelines for the Diagnosis and Treatment of Multiple Sclerosis (2023 Edition).

(2) Evidence of disease activity, meeting at least two of the following: (a) clinical relapse within the past 12 months confirmed by a neurologist; (b) MRI activity, including ≥1 new or enlarging T2 lesion or ≥1 new gadolinium-enhancing T1 lesion; (c) disability progression defined by an increase in EDSS score from baseline (≥1.0 point if baseline EDSS ≥1.0; ≥1.5 points if baseline EDSS = 0), sustained for ≥6 months and not attributable to a single relapse.

(3) Relapsed/refractory disease despite ≥12 months of disease-modifying therapy (DMT), including inadequate response, intolerance, contraindication, or relapse during or after treatment discontinuation.

4. Documented intolerance or inadequate response to prior therapy with glucocorticoids and at least two additional immunosuppressive or immunomodulatory agents, administered at effective doses for ≥3 months.

5. Adequate organ function, defined as:

(1) Hematologic: ANC ≥0.5 × 10^9/L; platelets ≥20 × 10^9/L; hemoglobin ≥60 g/L. (2) Coagulation: INR ≤1.5 × ULN and APTT ≤1.5 × ULN. (3) Hepatic: AST and ALT ≤5 × ULN; total bilirubin ≤1.5 × ULN. (4) Renal: serum creatinine ≤1.5 × ULN or creatinine clearance ≥30 mL/min (Cockcroft-Gault).

(5) Cardiac: NYHA class I-II; LVEF ≥50%; no pericardial effusion; and no clinically significant ECG abnormalities.

(6) Pulmonary: oxygen saturation ≥92% on room air; no clinically significant pleural effusion.

6. Estimated life expectancy greater than 6 months. 7. Agreement to use effective contraception throughout the treatment period and for 24 months after CAR T-cell infusion; women of childbearing potential must have a negative pregnancy test at screening.

8. Ability and willingness to provide written informed consent.

Exclusion Criteria:

1. Prior history of, or concurrent, other active malignancies, including malignancy-associated polymyositis/dermatomyositis. Exceptions include cervical carcinoma in situ, noninvasive basal cell or squamous cell skin cancer, localized prostate cancer treated with curative intent, or ductal carcinoma in situ after curative surgery, provided the participant is considered cured or has been disease-free for at least 2 years.

2.Severe pulmonary disease within the past 3 months, such as moderate-to-severe pulmonary arterial hypertension (mean pulmonary artery pressure >60 mmHg by echocardiography), requirement for supplemental oxygen via reservoir mask at screening, or requirement for noninvasive or invasive mechanical ventilation.

3.At screening, serum IgA, IgG, and IgM below the lower limit of normal (LLN). 4.Use of any of the following medications or therapies within the specified time windows:

1. Use of B-cell-depleting therapy within 1 month prior to screening and assessed by the investigator as not having failed therapy, including agents targeting CD19, CD20, CD22, CD52, CD38, or BCMA (monoclonal antibodies or bispecific antibodies).
2. High-dose intravenous human immunoglobulin (IVIG) within 1 month prior to screening.
3. Therapeutic-dose systemic corticosteroids within 24 hours prior to lymphodepleting conditioning (prednisone >20 mg/day or equivalent).
4. Corticosteroid pulse therapy within 2 weeks (defined as prednisone ≥500 mg/day or equivalent).
5. Telitacicept within 2 weeks prior to screening, or belimumab within 3 weeks prior to screening.

5. History of severe central nervous system (CNS) disease or related symptoms within the past 6 months (simple trigeminal neuralgia excluded), including but not limited to neuropsychiatric lupus, cerebrovascular disease, encephalitis, brain injury, aneurysm, cerebellar disease, organic brain syndrome, Parkinson's disease, as well as symptoms such as seizures/convulsions, aphasia, or dementia.

6. Lupus crisis within 3 months prior to screening, such as active CNS lupus, severe autoimmune hemolytic anemia, severe immune thrombocytopenic purpura, severe granulocytopenia, severe myocardial injury, severe lupus pneumonitis or pulmonary hemorrhage, severe lupus hepatitis, severe vasculitis, or other severe lupus manifestations.

7. Severe renal disease, including severe lupus nephritis within 8 weeks prior to screening (defined as urine protein >4 g/24 hours, or serum creatinine >1.5 × ULN, or creatinine clearance <30 mL/min by Cockcroft-Gault), active nephritis requiring use of protocol-prohibited medications, or nephritis requiring prednisone >500 mg/day (or equivalent systemic corticosteroids) for ≥14 days.

8.Severe hypersensitivity/allergy to any lymphodepleting conditioning agent used in this study or to any component related to CAR T-cell manufacture/culture.

9.Hepatitis B: positive HBsAg with detectable HBV DNA in peripheral blood;Hepatitis C: positive anti-HCV with detectable HCV RNA; Syphilis: RPR/TRUST titer ≥1:8; HIV: positive HIV antibody.

10.Uncontrolled fungal, bacterial, or viral infection, or any other infection that, in the investigator's judgment, makes the participant unsuitable for study participation.

11. History of major organ transplantation (e.g., heart or lung transplantation).

12. Active tuberculosis or latent tuberculosis at screening (defined as a positive tuberculin skin test or positive interferon-gamma release assay), regardless of the absence of clinical symptoms or imaging evidence.

13. Any of the following cardiovascular diseases within 6 months prior to screening, including but not limited to:

1. Congestive heart failure, myocardial infarction, unstable angina, coronary angioplasty, stent implantation, or coronary/peripheral artery bypass surgery.
2. Severe arrhythmias requiring treatment (e.g., sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes); congenital long QT syndrome; left anterior fascicular block (bifascicular block). Asymptomatic right bundle branch block is permitted.
3. Uncontrolled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg), or a history of hypertensive crisis or hypertensive encephalopathy.

14. History of other autoimmune diseases (other than the target indication) requiring systemic therapy, including but not limited to eosinophilic granulomatosis with polyangiitis, cryoglobulinemic vasculitis, inclusion body myositis, anti-glomerular basement membrane disease, Behçet's disease, or Takayasu arteritis.

15. Non-IIM myopathy, such as drug-induced myopathy, or a family history of human immunodeficiency virus (HIV)-associated myopathy.

16. Pregnancy or breastfeeding. 17. Receipt of a live vaccine within 6 weeks prior to lymphodepleting conditioning.

18. Participation in another interventional clinical study within 3 months prior to signing informed consent, receipt of an active investigational drug, or intention to participate in another clinical trial during this study period, or receipt of autoimmune disease treatment not specified in the protocol during the study period.

19. Psychiatric disorders such as depression with suicidal ideation or suicidal tendency.

20. Any other condition or factor that, in the investigator's judgment, makes the participant unsuitable for enrollment or may affect participation in or completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of participants with adverse events (AEs), serious adverse events (SAEs), laboratory abnormalities, and adverse events of special interest (AESIs: CRS and ICANS), graded per CTCAE v5.0 and ASTCT 2019 criteria | From Day 0 through Month 24 after infusion (including Day 1-28 observation and Month 2-24 follow-up).
  AEs will be collected from the time of signing the informed consent form through 2 years after CAR-T infusion or the exit visit, whichever occurs first; if disease relapse occurs within 6 months after infusion, AEs will be collected as much as possible through 6 months post-infusion with participant cooperation. All AEs will be coded using MedDRA and summarized by System Organ Class (SOC) and Preferred Term (PT) as the number and percentage of participants with events. AE severity will be summarized using CTCAE v5.0. CRS and ICANS will be summarized using ASTCT 2019 grading criteria. AESIs (including CRS and ICANS) and SAEs (including death) will be listed separately.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Boren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided